CLINICAL TRIAL: NCT02971306
Title: Granulocyte Colony Stimulating Factor Plus N-Acetyl Cysteine In Severe Alcoholic Hepatitis
Brief Title: G-CSF Plus NAC In Severe Alcoholic Hepatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-CSF and NAC in AH
Record Dates: First submitted 2016-11-09; First posted 2016-11-22 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Alcoholic Hepatitis
Keywords: alcoholic hepatitis; alcoholic liver disease; jaundice; ascites; regeneration
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Diseases, Alcoholic; Jaundice; Ascites | interventions — Granulocyte Colony-Stimulating Factor; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Medical therapy (Active Comparator): standard medical therapy
  Interventions: Drug: standard medical therapy
- G-CSF (Experimental): standard medical therapy plus G-CSF- 5μg/Kg s.c every 12 hours for 5 consecutive days
  Interventions: Drug: standard medical therapy; Drug: G-CSF
- G-CSF and NAC (Experimental): standard medical therapy plus G-CSF- 5μg/Kg s.c every 12 hours for 5 consecutive days plus NAC (day 1: NAC at 150, 50, and 100 mg/kg in 250, 500, and 1000 ml of 5% glucose solution over 30 minutes, 4 hours, and 16 hours, respectively; days 2 through 5: 100 mg/kg/day in 1000 ml of 5% glucose solution)
  Interventions: Drug: standard medical therapy; Drug: G-CSF; Drug: n-Acetylcysteine

INTERVENTIONS:
Drug: standard medical therapy — Standard medical therapy involves primary treatment with pentoxifylline at a dose of 400 mg three times a day and normal hospital nutrition (1800 to 2000 kcal per day). Diuretics, sodium restriction and albumin for treatment of ascites or fresh frozen plasma for coagulopathy or antibiotics for any focus of infection as spontaneous bacterial peritonitis (SBP), pneumonia, cellulitis, and urinary tract infection as indicated.
Drug: G-CSF — G-CSF- 5μg/Kg s.c every 12 hours for 5 consecutive days
  Arms: G-CSF; G-CSF and NAC
Drug: n-Acetylcysteine — n-Acetylcysteine at 150, 50, and 100 mg/kg in 250, 500, and 1000 ml of 5% glucose solution over 30 minutes, 4 hours, and 16 hours, respectively; days 2 through 5: 100 mg/kg/day in 1000 ml of 5% glucose solution
  Arms: G-CSF and NAC

SUMMARY:
Alcoholic hepatitis is related to very high mortality rate. About 40% of the patients are died within first 6 months after the detection of the clinical syndrome. Therefore, it is very essential for proper diagnosis and early treatment. In response to acute or chronic liver damage, bone marrow derived stem cells can spontaneously populate liver and differentiate into hepatic cells. Animal and human studies suggested that injured hepatocyte may be replaced by pluripotent bone marrow cells. However, this hepatocyte repopulation is highly dependent on varieties of liver injury and therapeutic conditions6. The studies has suggested Granulocyte-colony stimulating factors (G-CSF) can regenerate hepatocyte by fusing with hematopoietic cells, thereby enhancing the liver histology and survival rate.

G-CSF is a cytokine capable to regulate a number of functions in neutrophils. In three recent studies mobilization of bone marrow stem cells induced by G-CSF was observed in patients with alcoholic hepatitis. In two of this studies there was a survival benefit with the use of G-CSF.

Alcoholism leads to decrease in endogenous antioxidant potential. Alcoholic liver disease (ALD) patients show low endogenous antioxidants. Chronic ethanol consumption cause selective deficiency in the availability of reduced glutathione (GSH) in mitochondria has been reported. This is due to impaired functioning of GSH transporter from cytosol to mitochondrial matrix. The effect on glutathione replenishing potential by N-acetyl cysteine (NAC) can be used to reduce oxidative stress, which also has excellent safety profile. Therefore, NAC can be used for severe alcoholic hepatitis treatment due to its therapeutic potential factor. NAC also inhibit apoptosis and pro-inflammatory cytokine production. In a study high doses of intravenous N-acetyl cysteine therapy for 14 days conferred neither survival benefits nor early biological improvement in severe alcoholic hepatitis patients with adequate nutritional support.However, these results must be viewed with caution, since the study suffered from a lack of power. In a recent study, NAC and corticosteroids combination therapy benefits among patients with severe acute alcoholic hepatitis in 1 month survival, although the final outcome at 6 month survival was not improved. There are no studies on the use of combination therapy of NAC plus G-CSF in patient with severe alcoholic hepatitis.

Therefore we plan to study the safety and efficacy of combination therapy of G-CSF and NAC in the patients with alcoholic hepatitis.

DETAILED DESCRIPTION:
Patients with severe alcoholic hepatitis, admitted to Department of Hepatology PGIMER, Chandigarh from July 2014 to December 2016 will be included in the study.

METHODS

This will be an open label trial. A randomization code is generated by random number table. The patients will be randomized to receive standard medical therapy of pentoxifylline only as control and combination therapy of Pentoxifylline with NAC and G-CSF as cases. There will be one control and two cases as below:

1) Pentoxifylline (control) 2) Pentoxifylline+G-CSF (case 1) 3) Pentoxifylline+G-CSF +NAC (case2) A) Pentoxifylline 400 mg thrice daily for 28 days A) Pentoxifylline 400 mg thrice daily for 28 days plus G-CSF 5 mcg/kg every 12 hourly for consecutive 5 days A) Pentoxifylline 400 mg thrice daily for 28 days plus G-CSF 5 mcg/kg every 12 hourly for 5 days plus NAC 300 mg/kg on day 1 (150 mg/kg in 250 ml of 5% dextrose over a minute of 30 minutes,50 mg/kg in 500ml 5% dextrose over a period of 4 hours, 100mg /kg in 1000 ml of 5% dextrose over a period of 16 hours ) and on day 2 through 5 100mg /kg/day in 1000ml of glucose solution.

This will be a single time therapy. Patients will be admitted in the department of hepatology and will be assessed everyday clinically as well as by laboratory tests during therapy to assess safety and effects of treatment.

1. Total leukocytes count will be assessed daily.
2. Circulating CD 34 positive cells will be measured on day 0 and 6 of G-CSF therapy.
3. In addition, ultrasonography will be performed at day 1 and 6 in order to evaluate difference in spleen size and portal vein flow.
4. Biochemical, coagulation, and hematological parameters (Liver function tests, Renal Function Tests, Prothrombin Time, International Normalised Ratio, etc.) will be monitored periodically, daily for 1 week, then weekly for 1month and monthly for three month.

All patients will be followed at weekly interval for 1 month and then monthly for 3 months.

Outcome:

Primary Objectives:

Survival at 3 months

Secondary Objectives:

Mobilisation of CD34 positive cells in peripheral blood. Clinical/biochemical improvement in liver function profile. Improvement in prognostic scores-Maddrey's Discriminant function, MELD score, and Child score.

Safety and efficacy of G-CSF and NAC in alcoholic hepatitis

ELIGIBILITY:
Inclusion Criteria:

Alcoholic hepatitis patients:

1. More than 10 years of heavy alcohol consumption (mean intake ≈ 100 g/day).
2. Elevated aspartate aminotransferase level (but <500 IU per millilitre) and Ratio ofAST/ALT≥2 times
3. Elevated serum total bilirubin level ≥ 5 mgdL (86 μmol/L)
4. Elevated INR(≥1.5) and
5. Neutrophilia. Patient with Maddrey's DF of≥ 32 will be included in the study, with or without biopsy.

Exclusion Criteria:

1. Age < 18 and > 75 years
2. Hepatocellular carcinoma or portal vein thrombosis
3. Refusal to participate in the study
4. Serum creatinine >1.0 mg%
5. Hepatic encephalopathy- grade 3 or 4
6. Upper gastrointestinal bleed in last ten days
7. Uncontrolled bacterial infection
8. Human immunodeficiency virus, Hepatitis B virus, Hepatitis C virus seropositivity, Autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha1-antitrypsin deficiency
9. Pregnancy
10. Glucocorticoid treatment
11. Significant co-morbidity
12. Previous known hypersensitivity to G-CSF/NAC

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Primary end point- Survival at the end of 90 days | 90 days

SECONDARY OUTCOMES:
mobilization of CD34+ cells in peripheral blood | 6 days
improvement in MELD score | 90 days
Number of participants with treatment-related adverse events in the different treatment groups | 90 days
improvement in modified Discriminant Factor | 90 days
improvement in Child Turcotte Pugh score | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Hepatology, PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh V, Keisham A, Bhalla A, Sharma N, Agarwal R, Sharma R, Singh A. Efficacy of Granulocyte Colony-Stimulating Factor and N-Acetylcysteine Therapies in Patients With Severe Alcoholic Hepatitis. Clin Gastroenterol Hepatol. 2018 Oct;16(10):1650-1656.e2. doi: 10.1016/j.cgh.2018.01.040. Epub 2018 Jan 31. PMID 29391265